CLINICAL TRIAL: NCT04682964
Title: Bacteriophage Therapy in Acute Tonsillitis
Brief Title: Bacteriophage Therapy in Tonsillitis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tashkent State Medical University (Tashkent Pediatric Medical Institute), Uzbekistan (Other)
Responsible Party: Principal Investigator, Turdieva Shokhida Tolkunovna, MD, МD, associate professor of the Department "Outpatient care", Tashkent State Medical University (Tashkent Pediatric Medical Institute), Uzbekistan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TashkentPediatricMI
Record Dates: First submitted 2020-12-09; First posted 2020-12-24 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Acute Tonsillitis
Keywords: acute tonsillitis; children; bacteriophage; immunity; ambulatory treatment
MeSH Terms: interventions — Phage Therapy

STUDY DESIGN:
Intervention Model Description: Children aged 3 to 14 years with clinically diagnosed acute tonsillitis will receive bacteriophage therapy using a liquid pyobacteriophage complex (liquid pyobacteriophage complex - PCL).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nebulizer inhalation bacteriophage therapy (Experimental): To study the effects of bacteriophage therapy on acute tonsillitis in children and adolescents in an outpatient setting.
  Interventions: Drug: Nebulizer inhalation irrigation of the mucous membranes of the tonsils with a bacteriophage.

INTERVENTIONS:
Drug: Nebulizer inhalation irrigation of the mucous membranes of the tonsils with a bacteriophage. — Bacteriophage therapy using a liquid complex of pyobacteriophages (pyobacteriophage complex liquid - PСL). PСL was administered via nebulizer inhalation to irrigate the mucous membranes of the tonsils. In total, 5 ml of PCL was inhaled for up to 10 minutes once every 5 days.
  Other Names: Bacteriophage therapy.

SUMMARY:
The patients received bacteriophage therapy with a liquid piobacteriophage complex (liquid pyobacteriophage complex - PCL). PСL was administered via nebulizer inhalation to irrigate the tonsil mucosa. A total of 5 ml of PCL was inhaled for 10 minutes every 5 days. The drug causes the lysis of certain bacteria, including staphylococcus, enterococcus, streptococcus, enteropathogenic E. coli, Proteus vulgaris, Proteus mirabilis, Pseudomonas aeruginosa, Klebsiella pneumoniae and Klebsiella oxytoca. The choice of this drug was based on bacteriological studies.

DETAILED DESCRIPTION:
Comprehensive outpatient treatment was based on standard clinical guidelines, and symptomatic treatment was performed. On the first day of diagnosis, patients were prescribed complex antibacterial therapy on the basis of possible causative agents. Subsequently, antibiotic therapy was adjusted based on the results of the bacteriological examinations. A total of 67 patients received bacteriophage therapy using a liquid complex of pyobacteriophages (pyobacteriophage complex liquid - PСL). PСL was administered via nebulizer inhalation to irrigate the mucous membranes of the tonsils. In total, 5 ml of PCL was inhaled for up to 10 minutes once every 5 days.

The drug causes lysis of specific bacteria including Staphylococcus, Enterococcus, Streptococcus, enteropathogenic Escherichia coli, Proteus vulgaris, Proteus mirabilis, Pseudomonas aeruginosa, Klebsiella pneumoniae, and Klebsiella oxytoca. The drug is recommended for use for diseases of the ear, throat, nose, respiratory tract and lungs; inflammation of the sinuses and middle ear; tonsillitis; pharyngitis; laryngitis; tracheitis; bronchitis; pneumonia, pleurisy; and other inflammatory diseases. The choice of this drug was based on bacteriological studies.

ELIGIBILITY:
Inclusion Criteria:

* children from 3 to 14 years old.
* children with sore throat.
* children diagnosed with acute tonsillitis.
* children diagnosed with acute respiratory infection (rhinitis, sinusitis, nasopharyngitis).
* children with the opportunity to visit the outpatient clinic.
* children with the ability to receive inhalation therapy.
* children from parents (or guardians) who have given written permission to conduct clinical and laboratory research.

Exclusion Criteria:

* children under 3 years old and over 14 years old.
* children receiving hospital treatment.
* children with acute respiratory tract diseases (bronchitis, pneumonia, pleurisy).
* children with сhronic respiratory tract diseases (bronchitis, pneumonia).
* children who are allergic to antibiotics.
* children with cancer, immunological and hematological diseases.
* children with severe psychological illnesses (schizophrenia, mental retardation, etc.)
* children with cancer, immunological and hematological diseases.
* children with tuberculosis.

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical observation of sick children. | study of one patient - 4 weeks
  Children with clinically diagnosed acute tonsillitis are examined. The clinical study will be carried out on an outpatient basis in cooperation with the clinic of the Tashkent Pediatric Medical Institute. Prior to the study, written permission will be obtained from the parents or guardians of the children to participate in the study. Investigated: anamnesis of the child, the course of the disease, complaints of parents about the child's condition, body temperature in dynamics, visually - the state of the nasopharynx, the manifestation of clinical symptoms (sore throat, headaches, difficulty swallowing food, aphonia, and other signs) in dynamics, the functional state of internal organs (percussion, palpation and auscultation).
Laboratory research methods. | study of one patient - 2 weeks
  All examined children will undergo general clinical examination and pharyngoscopy. Additionally, all patients will have tonsil swabs for bacteriological examination (bacteriological culture, n x 10⁴/mL ) according to the standard technique. Also, swabs from the nasopharynx will be taken for viral lesions by the standard method - PCR (polymerase chain reaction). The research will be carried out in specialized laboratories.
Experimental clinical stage. Bacteriophage therapy. | study of one patient - 4 weeks
  Comprehensive outpatient treatment will be based on standard clinical guidelines. Patients will be prescribed antibiotic therapy based on possible pathogens. Patients will receive bacteriophage therapy using a liquid pyobacteriophage complex (liquid pyobacteriophage complex - PCL), through nebulizer inhalation to irrigate the mucous membranes of the tonsils. Just 5 ml PCL for 10 minutes once every 5 days. Efficacy will be studied based on immunological studies.A study of cellular (class of T-lymphocytes, Inflammatory cytokines (e.g., IL-1,2,4,5,6,11,13 - U/ml) and TNF-α) and humoral ( IgA / IgM / IgG -IU/mL) immunity in children will be carried out, using (Enzyme Linked Immunosorbent Assay) ELISA which is an immunoassay, suited to the determination of antibodies in the field of infectious serology.

SECONDARY OUTCOMES:
The second stage of the study (statistical). | 4 weeks
  The results will be analyzed using a statistical program based on Excel 2017 (Microsoft Office 2017). Clinical signs will be calculated as a percentage (%) incidence. We will calculate the chi-square (χ2) test or Fisher's exact test (for expected values <5) to assess if certain pairs of microbes are more common than expected by chance in bacteriological examination. In addition, we will use the Kruskal-Wallis test to compare the average delay between disease onset and sample collection between samples containing one or more organisms. When evaluating immunological analyzes, characterizing the statistical significance of differences, the Student's t-test will be used with the definition of the confidence interval. The X-square test will be used to assess the frequency of identifying qualitative features. In all analyzes, P ≤ 0.05 was considered significant.

CONTACTS AND LOCATIONS:
Overall Officials: Shokhida T. Turdieva, MD, Study Director — Tashkent State Medical University (Tashkent Pediatric Medical Institute), Uzbekistan
Locations (1):
- Tashkent Pediatric Medical Institute, Tashkent, Uzbekistan

IPD SHARING:
Plan to Share IPD: Yes
We are planning to create a joint project to research the treatment of bacterial infection in children with respiratory diseases by COVED-19.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2021-2024
Access Criteria: Children 0-17 years old, after being diagnosed with COVID-19, with a bacterial infection of the upper respiratory tract. We will work together with children's hospitals and research centers.